CLINICAL TRIAL: NCT02255955
Title: The Effect of Naproxen Sodium + Codeine, and Paracetamol+ Codeine on Postoperative Laminectomy Pain
Brief Title: Postoperative Analgesia in Laminectomy
Acronym: (PAL)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Reyhan Polat, Medical Doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pstoperative pain
Record Dates: First submitted 2014-09-27; First posted 2014-10-03 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Postoperative Pain; Postoperative Laminectomy Pain
Keywords: naproxen sodium codeine; paracetamol codeine; disk surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Naproxen; Codeine; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 550 mg naproxen sodium and 30mg codeine (Experimental): Preoperatively patients received oral naproxen sodium codeine, postop contramal infused by PCA, and postoperative contramal consumption, side effects pain intensity measured by VAS.
  Interventions: Drug: 550 mg naproxen sodium and 30mg codeine
- 300 mg paracetamol and 30 mg codeine (Active Comparator): Preoperatively patients received oral paracetamol codeine, postop contramal infused by PCA, and postoperative contramal consumption, side effects pain intensity measured by VAS.
  Interventions: Drug: 300 mg paracetamol and 30 mg codeine
- Placebo (Placebo Comparator): Preoperatively patients received oral placebo tablet, postop contramal infused by PCA, and postoperative contramal consumption, side effects pain intensity measured by VAS.
  Interventions: Drug: placebo tablet

INTERVENTIONS:
Drug: 550 mg naproxen sodium and 30mg codeine — Postoperative contramal consumption, pain intensity, side effects
  Other Names: Apranax plus
  Arms: 550 mg naproxen sodium and 30mg codeine
Drug: 300 mg paracetamol and 30 mg codeine — Postoperative contramal consumption, pain intensity, side effects
  Other Names: geralgine K
  Arms: 300 mg paracetamol and 30 mg codeine
Drug: placebo tablet — Postoperative contramal consumption, pain intensity, side effects
  Arms: Placebo

SUMMARY:
Compare the analgesic effects of naproxen sodium codeine, paracetamol codeine and placebo on postoperative pain and tramadol (Contramal) consumption during the first 24 hour after a lumbar disk surgery.

DETAILED DESCRIPTION:
Compare the analgesic effects of naproxen sodium codeine paracetamol codeine and placebo on postoperative pain intensity measured by the visual analogue scale, and evaluated tramadol consumption and related side effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) 1 or 2 status patients scheduled for an elective lumbar disc surgery

Exclusion Criteria:

* were known allergies to any of the drugs used in this study
* peptic ulcer disease
* hepatic and renal dysfunction,
* emergency surgery
* inability to provide informed consent

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Contramal consumption | Postoperative 24 hour
  To assess contramal consumption

SECONDARY OUTCOMES:
Side effects | postoperative 24 hour
  nausea and vomiting
Pain intensity | postoperative 24 hour
  To assess postoperative pain intensity by visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Reyhan Polat, MD, Principal Investigator — Ministry of Health